CLINICAL TRIAL: NCT04599348
Title: Treatment of CFS and Fibromyalgia With HRG 80 Red Ginseng
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Principal Investigator, Jacob Teitelbaum, Principal investigator, Practitioners Alliance Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-HRG80-2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia; CFS
Keywords: Ginseng
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Ginseng treatment (Experimental): People with CFS or Fibromyalgia will receive HRG 80 Red GInseng
  Interventions: Dietary Supplement: HRG 80 Red Ginseng

INTERVENTIONS:
Dietary Supplement: HRG 80 Red Ginseng — A unique form of ginseng with the high level of active ginseng components similar to those found in the wild ginseng used in earlier studies.

SUMMARY:
Will a unique form of ginseng be clinically helpful in those with chronic fatigue syndrome and fibromyalgia?

DETAILED DESCRIPTION:
Ginseng has been shown in earlier studies to help fatigue in a number of conditions. But because of overharvesting, most ginseng is no longer have optimal levels of the active ginsenosides. A new technique has been developed to restore the level of active ginseng components those found in the wild ginseng used in earlier studies. This is available in a form called HRG 80 Red Ginseng.

The study is an open pilot study to explore whether this treatment would be helpful for improving clinical function and symptomatology in chronic fatigue syndrome and fibromyalgia. Current clinical experience is suggesting that it may be.

ELIGIBILITY:
Inclusion Criteria:

1. be diagnosed with CFS and/or fibromyalgia
2. live in the United States 3 - be over 18 years of age

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Composite Visual analog scale of symptoms | 6 weeks
  Composite Score visual analog scale (0 - 30 Visual analog scale units , with 30 VAS units representing optimal function) of energy, cognition, and overall well-being. Each on a 0-10 scale with 10 being healthy. The units are the same for all 3 allowing them to be combined into a single composite total score. This total score (0-30 with 30 being the best outcome ) is the primary outcome measure

SECONDARY OUTCOMES:
VAS of pain and sleep | 6 weeks
  VAS of pain and sleep

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Teitelbaum, Principal Investigator — FFTF LLC
Locations (1):
- Kona Research Center, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No